CLINICAL TRIAL: NCT06355557
Title: Human vs Machine: a Randomised Controlled Trial Comparing Traditional In-person Instruction, Artificial Intelligence Versus Virtual Reality for Learning Basic Critical Care Echocardiography
Brief Title: Human vs Machine: a RCT Comparing Traditional In-person Instruction, AI Versus VR for Learning Basic CCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Lau Yie Hui, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DSRB 2023/00640
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound
Keywords: artificial intelligence, echocardiography, POCUS

STUDY DESIGN:
Intervention Model Description: 3-arm prospective randomised controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 22 medical students (AI) (Active Comparator): medical students randomised to this arm
  Interventions: Other: AI enabled ultrasound system for self-directed learning
- 22 medical students (Simulator) (Active Comparator): medical students randomised to this arm
  Interventions: Other: Simulator for self-directed learning
- 22 medical students (control) (Active Comparator): medical students randomised to this arm
  Interventions: Other: traditional with human instructors

INTERVENTIONS:
Other: AI enabled ultrasound system for self-directed learning — use of the AI enabled ultrasound system for self-directed learning
  Other Names: AI-enabled ultrasound system (Kosmos(TM))
  Arms: 22 medical students (AI)
Other: Simulator for self-directed learning — use of the simulator for self-directed learning
  Arms: 22 medical students (Simulator)
Other: traditional with human instructors — Medical students who are randomised to this arm
  Arms: 22 medical students (control)

SUMMARY:
The aim of the study is to investigate if hands-on training for basic CCE with virtual reality simulators or guided by artificial intelligence is non-inferior to training by an experienced instructor.

DETAILED DESCRIPTION:
Basic (Level 1) Critical care echocardiography (CCE) involves using an ultrasound device to qualitatively assess the heart at the bedside. It is increasingly being used at the bedside for diagnostics and screening of key differential diagnoses. Increasingly, CCE is being taught to more medical staff from many fields in medicine, including emergency medicine, anaesthesiology, intensive care medicine and even family medicine. There is a wealth of learning resources online but access to direct supervision by trainers and in-person courses is can be limited and costly. At the time of the study, one local medical school incorporated a lecture there is no credentialling pathway within local medical schools or institution. There has been increasing use of machine learning in medical imaging and deep learning algorithms are now able to guide image acquisition and allow novices with minimal training in echocardiography to obtain diagnostic-quality images. Artificial intelligence (AI) in echocardiography may improve image by novices. Ultrasound hardware that implement machine learning software in real-time can help with structure detection and identification, but more studies are needed to determine the extent that AI impacts learning.

ELIGIBILITY:
Inclusion Criteria:

* Medical students will have limited clinical exposure to critical care echocardiography
* above the age of 21 years

Exclusion Criteria:

* prior attendance of a critical care echocardiography courses or
* refusal to participate in the study or complete both hands on sessions

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-04 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in image acquisition and structure identification at the end of 3 months. | 3 months
  The images acquired during that timeframe will be scored using the validated Rapid Assessment of Competency in Echocardiography Scale. The experienced CCE trainer who will score the subject will be blinded to which arm of the study the subject is in

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
local PDPA and data sharing rules

REFERENCES:
- [Derived] Lau YH, Acharyya S, Wee CWL, Xu H, Saclolo RP, Cao K, Fong WK. Effectiveness of traditional, artificial intelligence-assisted, and virtual reality training modalities for focused cardiac ultrasound skill acquisition: a randomised controlled study. Ultrasound J. 2025 Nov 21;17(1):61. doi: 10.1186/s13089-025-00469-7. PMID 41269495